CLINICAL TRIAL: NCT06056713
Title: The Effect of Hand Massage on Fatigue in Women With Cancer Receiving Brachytherapy Treatment
Brief Title: Hand Massage on Fatigue With Cancer Receiving Brachytherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Efe Arslan, ErciyesU, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 815-795
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hand Massage
Keywords: Hand Massage; Fatigue; Brachytherapy
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Interventions (Experimental): Hand massage should be done for 10 minutes, 5 minutes for each hand, before each brachytherapy (3 times in total in the 1st, 2nd and 3rd sessions).
  Interventions: Behavioral: Hand Massage
- Control Group (No Intervention): The control group did not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: Hand Massage — The hand massage application lasted 10 minutes, 5 minutes on each hand, before each brachytherapy (3 times in total in the 1st, 2nd and 3rd sessions).
  Arms: Experimental Interventions

SUMMARY:
This randomized controlled trial was designed to examine the effect of hand massage on the level of fatigue in patients receiving BT therapy. Randomized controlled trial was conducted in the radioterapi outpatient clinic of university hospital located in a large city in Turkey. When 12 patients were included in each group, it was determined that the power was 90% at the 5% Type I error level, and a total of 24 women with gynecological cancer were included in the study. The primary outcome of this study was the mean difference in fatigue scores between the groups following the three brachtherapy cycles hand intervention. Patient Information Form and Brief Fatigue Inventory (BFI) used. This study predicted that hand massage applied in each session, starting from the first session of brachytherapy application, would reduce the level of fatigue in women.

DETAILED DESCRIPTION:
Therefore, this study aimed to compare the effects of hand massage intervention the level of fatigue in patients receiving BT therapy. . This randomized clinical trial was conducted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* underwent BT regularly
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Having skin problems
* with metastases,
* have bleeding or coagulation disorders,
* using complementary integrated therapy during the study,
* Having edema or wound in the hand area,
* not wanting to get a massage
* Patients receiving general anesthesia during the procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study was conducted in women with gynecological cancer
Enrollment: 24 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory (BFI) | The scale was filled in the baseline (after of the Hand massage).]
  The BFI, developed by Mendoza et al. (1999), was used to rapidly assess the severity and impact of cancer-related fatigue on daily living activities [33]. This inventory has nine items and measures fatigue severity (questions 1, 2, and 3) and fatigue interference in daily life activities (questions 4a, 4b, 4c, 4d, 4e, and 4f). Its reliability and validity, in the Turkish context, were determined by Usta Yeşilbalkan and Karadakovan (2005) and had a Cronbach's alpha value of Turkish version of 0.97 [34]. Each item of the BFI that consists of 9 items takes a value between 0-10 points.; higher scores indicate greater fatigue scores. Fatigue severity score is calculated by nine items and whereas fatigue interference score is calculated by summation of questions 4a, 4b, 4c, 4d, 4e, and 4f.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK EFE ARSLAN, PhD, Study Director — ERCİYES UNİVERSİTY
Locations (1):
- Dilek Efe Arslan, Kayseri, Melikgazi, Turkey (Türkiye)

REFERENCES:
- [Derived] Efe Arslan D, Kilic Akca N, Aslan D. The effect of hand massage on fatigue in women with cancer receiving brachytherapy: randomized clinical trial. Support Care Cancer. 2024 Dec 3;33(1):2. doi: 10.1007/s00520-024-09059-0. PMID 39625640